CLINICAL TRIAL: NCT07002840
Title: Effect of Engaging the Cross-legged Sitting in Rehabilitation Among Patients With Unilateral Hip Developmental Dysplasia According to Gait Parameters, Foot Pressure and Muscular Electrical Activity.
Brief Title: Effect of Cross-legged Sitting Among Patients With Unilateral Hip Developmental Dysplasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Hadeel Saad Alsirhani, Assistant Professor of Physical Therapy, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-13-S-(001)-(7371)
Record Dates: First submitted 2025-05-07; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Hip Developmental Dysplasia
Keywords: Rehabilitation; Gait; Foot pressure; Hip Developmental Dysplasia
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DDH kids who participated in rehabilitation programs with CLS (Experimental): The study sample includes kids with DDH who participated in rehabilitation programs with CLS.
  Interventions: Other: Cross- legged sitting position; Other: Physical Therapy Rehabilitation Program
- DDH kids who participated in usual rehabilitation programs without CLS (Active Comparator): The study sample includes kids with DDH who participated in rehabilitation programs without CLS.
  Interventions: Other: Physical Therapy Rehabilitation Program

INTERVENTIONS:
Other: Cross- legged sitting position — CLS in which the legs were crossed with hip and knee joints flexed
  Arms: DDH kids who participated in rehabilitation programs with CLS
Other: Physical Therapy Rehabilitation Program — Strengthening Exercises Stretching Exercises Range of Motion Exercises

SUMMARY:
One of the most common infant developmental diseases is Hip dysplasia which is mostly seen among female' babies and leads to hip instability due to partial or full hip dislocation [1]. Physical therapy's role plays a significant role in treating hip dysplasia by creating new walking habits as an adaptation way and compensation for the deformity [3]. Focusing on the muscles that produce hip abduction force is a basic item of the hip dysplasia rehabilitation program [4]. Cross-legged sitting position can be considered as a common and easy position that might enhance the range of motion of the lower limb joints [5].

While unilateral hip developmental dysplasia has been widely distributed among newborns, especially in the last few years, the role of engaging the cross-legged sitting technique as a part of physical therapy and rehabilitation programs on improving the temporospatial parameters, muscular electrical activity and foot pressure distributing is still not clear. Therefore, this study aimed to analyze the effects of engaging the cross-legged sitting technique as a part of physical therapy and rehabilitation program among patients with UHDD by comparing the group who participated in rehabilitation program with CLS to the other without.

To understand the importance of including Cross-legged sitting technique in physical therapy and rehabilitation program of Unilateral Hip Developmental Dysplasia (UHDD) to enhance the spatial and temporal measures, achieving a healthy distribution of foot pressure, increasing the electrical activity of lower limb muscles and improving the overall gait pattern.

No risks at all. All instruments and techniques in this study are safe and used regularly without any hazards.

The data will be stored and archived on a password-protected computer for safety and security purposes. After accomplishing the research and getting the outcomes, the results of the research may be published as an academic article in a peer-reviewed journal. In another word, no personal data will be published at all.

Taking part in the study and withdrawing at any time is completely voluntary with no need to give any reason.

ELIGIBILITY:
Inclusion Criteria:

* age group from 9 months to 10 years old
* all participants suffer from Unilateral Hip Developmental Dysplasia (UHDD)
* participants should be healthy in general

Exclusion Criteria:

Any participant with a history of neurological disorders, lower extremities previous surgical intervention, lower limb deformities, flat feet or high body mass index will be excluded from this study

Ages: 9 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-06-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Gait Temporospatial Parameters | 3 months
  Cadence will be measured by Gait Rite
Muscle Electrical Activity | 3 months
  Muscle Electrical Activity will be measured by Electromygraphy

SECONDARY OUTCOMES:
Foot Pressure | 3 months
  Average pressure will be measured using the foot pressure system

IPD SHARING:
Plan to Share IPD: No